CLINICAL TRIAL: NCT05507905
Title: Establishing the Optimal Frequency of Dance Movement for Neurocognitive and Physical Outcomes in People at Risk of Alzheimer's Disease
Brief Title: Effects of Dance and Music Appreciation on Brain Health and Fitness in People at Risk for Alzheimer's Disease
Acronym: IGROOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00086190; R01AG076669 (NIH)
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Risk; Aging; Dance
MeSH Terms: conditions — Alzheimer Disease | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: IGROOVE will randomize 200 participants meeting enrollment criteria in a 1:1:1:1 fashion to attend a music appreciation class or dance classes either 1x/week, 2x/week or 3x/week for 24 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dance 3 Times Weekly (3xD) (Experimental): Participants in this arm will attend classes 3 times a week for 24 weeks. During the 24 weeks, four different dance forms will be practiced. Each dance form will be taught for 6 weeks.
  Interventions: Behavioral: Dance Classes
- Dance 2 Times Weekly (2xD) (Experimental): Participants in this arm will attend classes 2 times a week for 24 weeks. During the 24 weeks, four different dance forms will be practiced. Each dance form will be taught for 6 weeks.
  Interventions: Behavioral: Dance Classes
- Dance 1 Time Weekly (1xD) (Experimental): Participants in this arm will attend a class 1 time a week for 24 weeks. During the 24 weeks, four different dance forms will be practiced. Each dance form will be taught for 6 weeks.
  Interventions: Behavioral: Dance Classes
- Music Appreciation Classes (MAC) (Active Comparator): In the MAC, the music associated with that dance form will be used as the subject for classes and will also change every 6 weeks.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — Music associated with dance forms in dance classes.
  Arms: Music Appreciation Classes (MAC)
Behavioral: Dance Classes — Four Different dance forms taught for 6 weeks each
  Arms: Dance 1 Time Weekly (1xD); Dance 2 Times Weekly (2xD); Dance 3 Times Weekly (3xD)

SUMMARY:
The purpose of this research study is to study the effects of dance movement and music on memory and cardiorespiratory fitness in older adults who are concerned about memory loss. The study aims to determine the optimal number of movement or music appreciation classes a week to support brain health and fitness. Participants will be people 62 years or older who are concerned about their memory, but do not yet have a diagnosis of cognitive impairment. If a participant is deemed qualified to participate, he/she will be placed into one of four groups and will attend 1, 2, or 3 group or music appreciation classes per week for 24 weeks (6 months). In addition to attending the group classes, participants will be asked to complete at least four study visits at Wake Forest Baptist Medical Center to complete various clinical assessments, including a brain MRI.

DETAILED DESCRIPTION:
IGROOVE is an individually randomized group treatment trial that is controlled and single-blind. It will enroll adults aged 62 years and older who are low-active, report a Cognitive Change Index score ≥16, do not meet criteria for mild cognitive impairment or dementia, are healthy enough to complete repeated graded exercise testing (GXT), and have no contraindications for magnetic resonance imaging (MRI). Randomization will be assessed to ensure equal distribution across study arms for these sex and body mass index (BMI) and will be stratified if necessary. New participants will be rolled into the intervention every 6 weeks. Data collection will take place at Atrium Wake Forest Baptist Health. Interventions will consist of dance classes or music appreciation classes designed and taught by local experts, and will take place in community sites, such as local dance studios, community centers, community gyms or churches. All intervention sites selected will be handicap accessible, well-lit, have appropriate flooring for safe dance movement, and access to sturdy chairs without wheels or arms.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive Change Index score ≥16
* Montreal Cognitive Assessment (MoCA) score ≥21
* Cognitively normal
* Low-active for past 6 months (<30 min, 3 days/week of exercise, including walking for exercise)
* MRI compatible
* Willing and able to complete exercise testing.
* Has reliable transportation or is able to use transportation provided by the study.
* English speaking (needed for group class participation)

Exclusion Criteria:

* Unable or unwilling to attend intervention classes 1-3x/week
* Current diagnosis of a major neurological disorder (Alzheimer's disease, Lewy body dementia, Frontotemporal dementia, Parkinson's disease, amyotrophic lateral sclerosis, etc.)
* Unwilling or unable to provide consent for study participation.
* Currently symptomatic or cortical stroke or stroke deemed exclusionary by the study physician. Reported or observed evidence of strokes on MRI will be reviewed on a case-by-case basis by the study physician to assess factors such as location, size, time since stroke, and residual symptoms.
* Taking medication during the intervention times that could negatively influence safety
* Current cancer treatment or other major medical problems that might independently affect cognition or movement or interfere with ability to attend intervention or study visits.
* Chronic vertigo.
* Enrolled in another interventional research study ≤3 months prior to beginning this study.
* Hip fracture, hip or knee replacement, or spinal surgery in past 6 months.
* Health contraindications for completing a graded exercise test and movement intervention, including uncontrolled hypertension (BP>200/110 mmHg), hypertriglyceridemia (TG>400 mg/dl), uncontrolled diabetes (HbA1c > 7.5), clinical evidence of anemia.
* Self-reports regularly drinking > 14 alcoholic beverages a week or current illicit drug use.
* Unable or unwilling to understand study procedures and comply with them for the duration of the study.

Min Age: 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen Consumption (VO2) | Baseline
  Assessed with Graded Exercise Test (GXT) Peak oxygen consumption, a marker of cardiorespiratory fitness (ml/kg/min) Shows effect on Cardio Respiratory Function.
Peak Oxygen Consumption (VO2) | Month 1
  Assessed with Graded Exercise Test (GXT) Peak oxygen consumption, a marker of cardiorespiratory fitness (ml/kg/min) Shows effect on Cardio Respiratory Function.
Peak Oxygen Consumption (VO2) | Month 3
  Assessed with Graded Exercise Test (GXT) Peak oxygen consumption, a marker of cardiorespiratory fitness (ml/kg/min) Shows effect on Cardio Respiratory Function.
Peak Oxygen Consumption (VO2) | Month 6
  Assessed with Graded Exercise Test (GXT) Peak oxygen consumption, a marker of cardiorespiratory fitness (ml/kg/min) Shows effect on Cardio Respiratory Function.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline
  Shows effect on Cognitive Function. Overall score from the RBANS; Average/Mild Impairment (standard scores of 70 or above), Moderate Impairment (standard scores from 55 to 69), and Severe Impairment (standard scores <54) Scores range from 40 to 160.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Month 1
  Shows effect on Cognitive Function. Overall score from the RBANS; Average/Mild Impairment (standard scores of 70 or above), Moderate Impairment (standard scores from 55 to 69), and Severe Impairment (standard scores <54) Scores range from 40 to 160.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Month 3
  Shows effect on Cognitive Function. Overall score from the RBANS; Average/Mild Impairment (standard scores of 70 or above), Moderate Impairment (standard scores from 55 to 69), and Severe Impairment (standard scores <54) Scores range from 40 to 160.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Month 6
  Shows effect on Cognitive Function. Overall score from the RBANS; Average/Mild Impairment (standard scores of 70 or above), Moderate Impairment (standard scores from 55 to 69), and Severe Impairment (standard scores <54) Scores range from 40 to 160.

SECONDARY OUTCOMES:
Class Attendance | Week 24
  Percent attendance (number of classes attended divided by number of classes offered in that arm)
Exercise Self-Efficacy | Baseline, Month 1, Month 3, Month 6
  Questionnaire that shows perceived confidence to engage in sufficient physical activity through accumulation over extended periods of time. The scale has a range of scores from 0-90. A higher number on the score represents a higher self-efficacy for exercise.

OTHER OUTCOMES:
Expanded short physical performance battery (eSPPB) | Baseline, Month 1, Month 3, Month 6
  The eSPPB is a brief test of global mobility function with excellent test-retest and inter-examiner reliability; is sensitive to change; is safe, and is a robust predictor of future physical disability and death. To avoid ceiling effects, investigators will use an expanded version (eSPPB) that increases the difficulty of the standing balance task by asking participants to hold postures for 30 instead of 10 seconds, adds a one-leg stand, and adds a narrow walk. The resulting score is normally distributed, continuous, and shows greater sensitivity to change. Dementia patients have lower scores on the SPPB so a favorable outcome for this outcome measure would be a significantly higher score post treatment. The eSPPB is scored as a continuous measure with a maximum score of 3.0 where 3 is the best possible outcome.
Gait Variability | Baseline, Month 1, Month 3, Month 6
  Assessed over 4m 3 times at usual pace and 3 times at fast pace using an instrumented mat (GAITRite System); it will provide data on the variability in these measures
Postural Sway | Baseline, Month 1, Month 3, Month 6
  Center of pressure (millimeter squared) collected using an Advanced Mechanical Technology Incorporated (AMTI) AccuSway biomechanics force platform.
Timed Up and Go (TUG) | Baseline, Month 1, Month 3, Month 6
  The Timed Up and Go test is used to assess a person's mobility and requires both static and dynamic balance. Time in seconds that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.
Overall physical activity | Baseline, Month 1, Month 3, and Month 6
  Overall volumes of movement in minutes per day
Dance Self-Efficacy | Baseline, Month 1, Month 3, Month 6
  For dance arms only. Perceived confidence to engage in an individual's specific dance program over extended periods of time. Five items scored on a scale of 0-10. A total score will be generated by summing scores from all five items and dividing by 5, for a potential range of total scores from 0-10, where a higher score is better.
Brief Psychological Needs Satisfaction and Frustration Scale (BPNSFS)--Satisfaction | Baseline, Month 1, Month 3, Month 6
  The BPNSFS yields overall scores on two scales: satisfaction and frustration. An overall score for satisfaction (total possible = 60, higher score is better) will be calculated.
Brief Psychological Needs Satisfaction and Frustration Scale (BPNSFS)--Frustration | Baseline, Month 1, Month 3, Month 6
  The BPNSFS yields overall scores on two scales: satisfaction and frustration. . An overall score for frustration (total possible = 60, lower score is better) will be calculated.
Magnetic Resonance Imaging (MRI)-Neuro imaging | Baseline, Month 6
  Grey matter volume (cm3); voxelwise freewater calculated from neurite orientation dispersion and density imaging (NODDI) image; from functional MRI (fMRI) graph theory analysis, global efficiency and modular structure
Average Heart Rate | Weekly up through Week 24
  Collected with chest-worn strap (beats per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hugenschmidt, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No